CLINICAL TRIAL: NCT02678559
Title: Preload Dependency Evaluation With Stroke Volume Variation During Alveolar Recruitment Manoeuvres
Acronym: PreDeARM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: CHU-0254
Record Dates: First submitted 2016-01-15; First posted 2016-02-10 (Estimated); Last update posted 2017-04-20 (Actual); Status verified 2017-04

CONDITIONS: Coronary Artery Disease; Coronary Artery Bypass; Hypovolemia; Anesthesia, General; Pulmonary Atelectasis
Keywords: Alveolar recruitment manoeuvre; Lung recruitment; Preload dependency; Cardiac surgery; Transoesophageal echocardiography
MeSH Terms: conditions — Coronary Artery Disease; Hypovolemia; Pulmonary Atelectasis

ARMS (2):
- TEE monitory system (Experimental): comparison between TEE and mini-invasive monitoring systems in accuracy of measurement of stroke volume variation during ARM.
  Interventions: Other: tee measurement; Other: flotrac measurement; Other: clearsight measurement
- mini-invasive monitoring system (Experimental): comparison between TEE and mini-invasive monitoring systems in accuracy of measurement of stroke volume variation during ARM.
  Interventions: Other: tee measurement; Other: flotrac measurement; Other: clearsight measurement

INTERVENTIONS:
Other: tee measurement
Other: flotrac measurement
Other: clearsight measurement

SUMMARY:
The principal aim is to assess impact of alveolar recruitment manoeuvres (ARM) on stroke volume variation, evaluated by trans-oesophageal echocardiography (TEE). These variations will be measured on preload dependency or preload independency status. The principal purpose is to determine if variations of stroke volume during standardized ARM can predict the preload dependency status.

DETAILED DESCRIPTION:
Population studied: anesthetized patients for cardiac surgery of coronary bypass.

Secondary endpoints : - comparison between TEE and mini-invasive monitoring systems in accuracy of measurement of stroke volume variation during ARM. These mini-invasive systems are : Clearsight system (Edwards Lifescience) and Flotrac system (Edwards Lifescience)

- Difference between pre and post-cardiopulmonary bypass status on principal purpose evaluation

ELIGIBILITY:
Inclusion Criteria:

* Adult patient Undergoing a surgical procedure of coronary artery bypass, with cardiopulmonary bypass Written consent collected

Exclusion Criteria:

* Emergency case
* Pericardial effusion
* Aortic or mitral valvulopathy
* Contraindication for : TEE, alveolar recruitment manoeuvre (emphysema, pneumothorax, hemodynamic instability), Ringer Lactate solution infusion
* Bad echogenicity
* Patient refusal to participate to the study
* No health insurance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Variation of stroke volume | at the beginning of cardiac surgery
  Variation of stroke volume measured by TEE, induced by a standardized ARM, at the beginning of cardiac surgery

SECONDARY OUTCOMES:
Velocity time integral (cm) | at the begining of cardiac surgery
  Velocity time integral (cm) (TEE measurement)
Velocity time integral (cm) | After fluid challenges until patient is on a preload independency state.
  Velocity time integral (cm) (TEE measurement)
Velocity time integral (cm) | After the cardiopulmonary bypass period, when sternotomy will be closed
  Velocity time integral (cm) (TEE measurement)
Cardiac index (l/min/m2) | at the begining of cardiac surgery
  Cardiac index (l/min/m2) (TEE measurement)
Cardiac index (l/min/m2) | After fluid challenges until patient is on a preload independency state.
  Cardiac index (l/min/m2) (TEE measurement)
Cardiac index (l/min/m2) | After the cardiopulmonary bypass period, when sternotomy will be closed
  Cardiac index (l/min/m2) (TEE measurement)
Right ventricle diameter/left ventricle diameter ratio | at the begining of cardiac surgery
  Right ventricle diameter/left ventricle diameter ratio (TEE measurement),
Right ventricle diameter/left ventricle diameter ratio | After fluid challenges until patient is on a preload independency state.
  Right ventricle diameter/left ventricle diameter ratio (TEE measurement),
Right ventricle diameter/left ventricle diameter ratio | After the cardiopulmonary bypass period, when sternotomy will be closed
  Right ventricle diameter/left ventricle diameter ratio (TEE measurement),
E/A ratio | at the begining of cardiac surgery
  E/A ratio (TEE measurement)
E/A ratio | After fluid challenges until patient is on a preload independency state.
  E/A ratio (TEE measurement)
E/A ratio | After the cardiopulmonary bypass period, when sternotomy will be closed
  E/A ratio (TEE measurement)
Sus-hepatic vein Doppler profile | at the begining of cardiac surgery
  Sus-hepatic vein Doppler profile (TEE measurement)
Sus-hepatic vein Doppler profile | After fluid challenges until patient is on a preload independency state.
  Sus-hepatic vein Doppler profile (TEE measurement)
Sus-hepatic vein Doppler profile | After the cardiopulmonary bypass period, when sternotomy will be closed
  Sus-hepatic vein Doppler profile (TEE measurement)
Invasive arterial pressure (mmHg) | at the begining of cardiac surgery
Invasive arterial pressure (mmHg) | After fluid challenges until patient is on a preload independency state.
Invasive arterial pressure (mmHg) | After the cardiopulmonary bypass period, when sternotomy will be closed
Heart rate (pulse/min) | at the begining of cardiac surgery
Heart rate (pulse/min) | After fluid challenges until patient is on a preload independency state.
Heart rate (pulse/min) | After the cardiopulmonary bypass period, when sternotomy will be closed
Expired CO2 (mmHg) | at the begining of cardiac surgery
Expired CO2 (mmHg) | After fluid challenges until patient is on a preload independency state.
Expired CO2 (mmHg) | After the cardiopulmonary bypass period, when sternotomy will be closed
Central venous pressure (mmHg) | at the begining of cardiac surgery
Central venous pressure (mmHg) | After fluid challenges until patient is on a preload independency state.
Central venous pressure (mmHg) | After the cardiopulmonary bypass period, when sternotomy will be closed
Pulse pressure variation (%) | at the begining of cardiac surgery
Pulse pressure variation (%) | After fluid challenges until patient is on a preload independency state.
Pulse pressure variation (%) | After the cardiopulmonary bypass period, when sternotomy will be closed
Perfusion index (pulsoxymeter) | at the begining of cardiac surgery
Perfusion index (pulsoxymeter) | After fluid challenges until patient is on a preload independency state.
Perfusion index (pulsoxymeter) | After the cardiopulmonary bypass period, when sternotomy will be closed
Stroke volume (ml) (Flotrac measurement) | at the begining of cardiac surgery
Stroke volume (ml) (Flotrac measurement) | After fluid challenges until patient is on a preload independency state.
Stroke volume (ml) (Flotrac measurement) | After the cardiopulmonary bypass period, when sternotomy will be closed
Stroke volume variation (%) (Flotrac measurement) | at the begining of cardiac surgery
Stroke volume variation (%) (Flotrac measurement) | After fluid challenges until patient is on a preload independency state.
Stroke volume variation (%) (Flotrac measurement) | After the cardiopulmonary bypass period, when sternotomy will be closed
Cardiac index (l/min/m2) (Flotrac measurement) | at the begining of cardiac surgery
Cardiac index (l/min/m2) (Flotrac measurement) | After fluid challenges until patient is on a preload independency state.
Cardiac index (l/min/m2) (Flotrac measurement) | After the cardiopulmonary bypass period, when sternotomy will be closed
Pulse pressure variation (%) (Flotrac measurement) | at the begining of cardiac surgery
Pulse pressure variation (%) (Flotrac measurement) | After fluid challenges until patient is on a preload independency state.
Pulse pressure variation (%) (Flotrac measurement) | After the cardiopulmonary bypass period, when sternotomy will be closed
Arterial pressure (mmHg) (Flotrac measurement) | at the begining of cardiac surgery
Arterial pressure (mmHg) (Flotrac measurement) | After fluid challenges until patient is on a preload independency state.
Arterial pressure (mmHg) (Flotrac measurement) | After the cardiopulmonary bypass period, when sternotomy will be closed
Stroke volume (ml) (Clearsight measurement) | at the begining of cardiac surgery
Stroke volume (ml) (Clearsight measurement) | After fluid challenges until patient is on a preload independency state.
Stroke volume (ml) (Clearsight measurement) | After the cardiopulmonary bypass period, when sternotomy will be closed
Stroke volume variation (%) (Clearsight measurement) | at the begining of cardiac surgery
Stroke volume variation (%) (Clearsight measurement) | After fluid challenges until patient is on a preload independency state.
Stroke volume variation (%) (Clearsight measurement) | After the cardiopulmonary bypass period, when sternotomy will be closed
Cardiac index (l/min/m2) (Clearsight measurement) | at the begining of cardiac surgery
Cardiac index (l/min/m2) (Clearsight measurement) | After fluid challenges until patient is on a preload independency state.
Cardiac index (l/min/m2) (Clearsight measurement) | After the cardiopulmonary bypass period, when sternotomy will be closed
Pulse pressure variation (%) (Clearsight measurement) | at the begining of cardiac surgery
Pulse pressure variation (%) (Clearsight measurement) | After fluid challenges until patient is on a preload independency state.
Pulse pressure variation (%) (Clearsight measurement) | After the cardiopulmonary bypass period, when sternotomy will be closed
Arterial pressure (mmHg) (Clearsight measurement) | at the begining of cardiac surgery
Arterial pressure (mmHg) (Clearsight measurement) | After fluid challenges until patient is on a preload independency state.
Arterial pressure (mmHg) (Clearsight measurement) | After the cardiopulmonary bypass period, when sternotomy will be closed
Near infrared spectroscopy : Cerebral SrO2 | at the begining of cardiac surgery
Near infrared spectroscopy : Cerebral SrO2 | After fluid challenges until patient is on a preload independency state.
Near infrared spectroscopy : Cerebral SrO2 | After the cardiopulmonary bypass period, when sternotomy will be closed

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France